CLINICAL TRIAL: NCT02509377
Title: Fetal Myelomeningocele Repair With Maternal BMI Between 35.0 and 40.0
Acronym: MOMSto40BMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24890
Record Dates: First submitted 2015-07-23; First posted 2015-07-28 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2017-06

CONDITIONS: Myelomeningocele; Pregnancy
Keywords: Fetal Surgery; Open Fetal Surgery; Elevated BMI; Body Mass Index; Spina Bifida
MeSH Terms: conditions — Meningomyelocele; Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMI 35.0 to 40.0 (Experimental): Mothers who meet all inclusion exclusion criteria for open fetal repair of myelomeningocele except BMI.
  These mothers have a BMI between 35.0 and 40.0
  Interventions: Procedure: Open Fetal Repair of Myelomeningocele

INTERVENTIONS:
Procedure: Open Fetal Repair of Myelomeningocele — Open Fetal Repair of Myelomeningocele when mothers BMI is elevated

SUMMARY:
Inclusion and exclusion criteria for fetal repair of MMC was established by the Management of Myelomeningocele Study (MOMS Trial) and these criteria are the standard of care throughout the United States. These criteria state exclusion for hypertension and diabetes which are known co-morbidities for obesity. Investigators plan to expand one exclusion criteria for open fetal repair surgery. Currently, an exclusion factor is a maternal BMI of 35.0 and greater.Investigators will maintain all other inclusion and exclusion criteria (including excluding for hypertension and diabetes) with the exception of expanding the BMI to include mothers with a BMI of 35.0 to 40.0. Co-morbidities of the research group will be compared to the comorbidities of the mothers published in the MOMS trial.

DETAILED DESCRIPTION:
The MOMS trial proved prenatal repair of myelomeningocele was an advantage over postnatal repair for the fetus/neonate/child and is the standard of care for maternal/fetal dyads who meet the inclusion exclusion criteria. Investigators plan to maintain all inclusion exclusion criteria for open fetal repair surgery of myelomeningocele with one exception, the expansion of the maternal BMI to 40.0. This population of mothers with a BMI of 35.0 to 40.0 have not been studied. The morbidities of these mothers will be compared to morbidities of mothers with a BMI less than or equal to 34.9 currently in the scientific literature.

ELIGIBILITY:
Inclusion Criteria:

* Maternal BMI 35.0 to 40.0
* No maternal documented co-morbidities
* Fetal MMC begins between thoracic 1 and sacral 1, on the spinal column.
* Evidence of fetal hindbrain herniation (hindbrain is being pulled down the spinal column).
* A gestational age is between 19 weeks 0 days and 26 weeks with evidence of placental membrane fusion.
* Documented normal fetal karyotype.

Exclusion Criteria:

* History of maternal alloimmunization problem
* Kell sensitization
* Risk of preterm birth
* History of spontaneous preterm birth
* Cervix <20mm in length
* Presence of cerclage
* Placental problem
* History of placental abruption
* Placental Previa
* Body-mass index of 40.1 or more
* Maternal contraindication to surgery
* Insulin-dependent pregestational diabetes
* Hypertension or preeclampsia
* HIV, hepatitis-B, or hepatitis-C positive
* Other medical condition of risk to mother
* Uterine problem
* Previous hysterotomy in the active uterine segment
* Severe fibroids
* Uterine malformation (bicornuate, arcuate, unicornuate, didelphys)
* No support person for periprocedural period
* Inadequate support at home for pregnancy
* Inadequate understanding of risks and benefits of fetal surgery
* Inability to comply with medical restrictions, follow up after fetal surgery
* Multiple gestation pregnancy (twins, triplets, etc.)
* A fetal anomaly unrelated to myelomeningocele (heart defect, lung lesions)
* Severe fetal kyphosis >30 degrees (curvature of the back)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Co-morbidities in mothers having fetal MMC repair | up to 40 weeks
  Measure the co-morbidity of mothers with a BMI of 35.0 to 40.0. Compare to published data in the MOMS trial.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Vlastos, Associate Professor, Principal Investigator — St. Louis University
Locations (1):
- SSM Cardinal Glennon Fetal Care Institute, St Louis, Missouri, United States

REFERENCES:
- [Result] Adzick NS, Thom EA, Spong CY, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Dabrowiak ME, Sutton LN, Gupta N, Tulipan NB, D'Alton ME, Farmer DL; MOMS Investigators. A randomized trial of prenatal versus postnatal repair of myelomeningocele. N Engl J Med. 2011 Mar 17;364(11):993-1004. doi: 10.1056/NEJMoa1014379. Epub 2011 Feb 9. PMID 21306277